CLINICAL TRIAL: NCT03511105
Title: A Randomised, Placebo-controlled, Double-blind (Sponsor Open), Segmental LPS Challenge Study to Investigate the Pharmacodynamics of GSK2798745 in Healthy Participants
Brief Title: Effects of GSK2798745 on Alveolar Barrier Disruption in a Segmental Lipopolysaccharide (LPS) Challenge Model
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to low probability of achieving a positive outcome on the primary endpoint.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 207464; 2017-002388-16 (EudraCT Number)
Record Dates: First submitted 2018-04-24; First posted 2018-04-27 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers
Keywords: Lipopolysaccharide; Pharmacodynamics; Healthy subjects; GSK2798745; Placebo; Segmental challenge
MeSH Terms: interventions — GSK2798745; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a randomised, placebo-controlled, parallel-group study wherein, subjects will be randomised in a ratio of 1:1 to receive 2 single doses of either 4.8 milligrams GSK2798745, then 2.4 milligrams GSK2798745 12 hours later; or a dose of placebo, then another dose of placebo 12 hours later.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This will be a double blind study where investigator, sub-investigators, other site staff and the subject will be blinded. Selected sponsor study team members will be unblinded to perform the interim analysis. This may include the medical monitor, study statistician, study programmer (and delegates) and study pharmacokineticist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects receiving GSK2798745 (Experimental): Eligible subjects will receive two tablets of 2.4 milligrams GSK2798745 on the morning of Day 1. Subjects will then undergo segmental challenge at 2 hours after first dose wherein LPS will be instilled into the right middle segment and saline control into the lingula segment of the contralateral side. The second dose of a single tablet of 2.4 milligrams of GSK2798745 will be administered 10 hours after LPS and saline challenge.
  Interventions: Drug: GSK2798745; Drug: Lipoplysaccharide from Escherichia Coli; Drug: Saline
- Subjects receiving matching Placebo (Placebo Comparator): Eligible subjects will receive two tablets of placebo on the morning of Day 1. Subjects will then undergo segmental challenge at 2 hours after first dose wherein LPS will be instilled into the right middle segment and saline control into the lingula segment of the contralateral side. The second dose placebo will be administered 10 hours after LPS and saline challenge.
  Interventions: Drug: Placebo; Drug: Lipoplysaccharide from Escherichia Coli; Drug: Saline

INTERVENTIONS:
Drug: GSK2798745 — GSK2798745 will be available as white to slightly colored, round biconvex tablets to be administered via the oral route.
  Arms: Subjects receiving GSK2798745
Drug: Placebo — Placebo matching to GSK2798745 will be available as white to slightly colored, round biconvex tablet to be administered via the oral route.
  Arms: Subjects receiving matching Placebo
Drug: Lipoplysaccharide from Escherichia Coli — LPS will be used as challenge agent. About 4 nanogram per kilogram of LPS will be instilled into the right middle lung segment via bronchoscopy 2 hours after dosing with GSK2798745 or placebo on Day 1.
Drug: Saline — Sterile saline (0.9%) will be used as control challenge. Saline will be instilled into the lingula segment of contralateral side of lung via bronchoscopy 2 hours after dosing with GSK2798745 or placebo on Day 1.

SUMMARY:
The primary objective of the study is to investigate the effect of GSK2798745 on alveolar-septal barrier permeability following LPS challenge in healthy subjects. The influx of protein-rich fluid into the lung due to damage to the alveolar capillary barrier, with resultant adverse effects on respiratory function, is a fundamental underlying defect in Acute Respiratory Distress Syndrome (ARDS). In this Phase 1, proof-of-mechanism study, a LPS challenge will be used as a surrogate injury model to investigate the effects of Transient receptor potential vanilloid 4 (TRPV4) channel blockade on alveolar-septal barrier permeability in man. This is a randomised, placebo-controlled, parallel group, double-blind (sponsor-open), segmental LPS challenge study of GSK2798745 in healthy subjects. Subjects will be randomised in a ratio of 1:1 to take 2 single doses of either 4.8 milligrams GSK2798745 followed by 2.4 milligrams GSK2798745 after 12 hours or a dose of placebo followed by another dose of placebo after 12 hours. The first dose will be administered on Day 1 at 2 hours before Baseline bronchoalveolar lavage (BAL) sampling from a segment in the left lower lobe of lung. LPS 4 nanogram per kilogram will subsequently be instilled into the right middle segment and saline control into the lingula segment of the contralateral side. The second dose of study treatment will be administered 10 hours after LPS challenge followed by post-dose BAL sampling on Day 2. Each subject will take approximately 5 weeks to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests (including a normal coagulation profile), ECGs, vital signs and spirometry. In the event of out-of-range results of safety tests, the tests may be repeated once within the screening window. If a retest result is again outside the reference range and considered clinically significant by the investigator and GlaxoSmithKline (GSK) medical monitor, the subject will be considered a screen failure.
* Normal spirometry (FEV1 >=80% of predicted, FEV1/FVC ratio >=70%) at Screening and before dosing.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 19 to 29.9 kilogram per square meter (kg/m^2)(inclusive).
* A male subject must agree to use contraception during the treatment period and for at least 7 days after the last dose of study treatment and refrain from donating sperm during this period.
* A female is eligible to participate if she is not of childbearing potential.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.

Exclusion Criteria:

* Significant history of or current cardiovascular, respiratory (e.g., asthma, chronic obstructive pulmonary disorder (COPD), bronchiectasis, active Tuberculosis [TB]), hepatic, renal, gastrointestinal, endocrine, hematological, autoimmune or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Subject who, in the investigator/designee's judgement, poses a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behavior and/or any evidence of suicidal ideation on any questionnaires e.g., Type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) in the last 5 years.
* Active ulcer disease or gastrointestinal bleeding at the time of Screening (positive FOBT at Screening).
* Abnormal blood pressure as determined by the investigator.
* Alanine aminotransferase (ALT) or bilirubin >1.5 times upper limit of normal (ULN) (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according Fridericia's formula (QTcF) >450 milliseconds (msec).
* At risk of Torsades de pointes (e.g., a personal history or a family history of sudden unexplained death, long QT, familial cardiac syndrome, or cardiomyopathy).
* Chronic or acute infection within the 4 weeks before dosing, (e.g., upper and lower respiratory infection within the 4 weeks before dosing).
* Major (as per investigator judgment) surgery within the last 12 weeks prior to randomisation or planned within 3 months of Screening.
* Use of prescription or non-prescription drugs (except paracetamol), including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) before the first dose of study medication, unless, in the opinion of the investigator and GSK Medical Monitor, the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator and/or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliters (mL) within 3 months.
* The subject has participated in a clinical trial and has received an investigational product within the following time period before the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months before the first dosing day.
* Presence of hepatitis B surface antigen (HBsAg) at Screening.
* Positive hepatitis C antibody test result at Screening. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C Ribonucleic acid (RNA) test is obtained.
* Positive Hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment. Test is optional and subjects with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.
* A positive pre-study drug/alcohol/cotinine screen.
* A positive test for immunodeficiency virus (HIV) antibody.
* Regular use of known drugs of abuse.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Current smoker or a history of smoking within 6 months of screening, or a total pack year history of >5 pack years. [number of pack years = (number of cigarettes per day/20) x number of years smoked].

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20768

REFERENCES:
- [Background] Mole S, Harry A, Fowler A, Hotee S, Warburton J, Waite S, Beerahee M, Behm DJ, Badorrek P, Muller M, Faulenbach C, Lazaar AL, Hohlfeld JM. Investigating the effect of TRPV4 inhibition on pulmonary-vascular barrier permeability following segmental endotoxin challenge. Pulm Pharmacol Ther. 2020 Oct;64:101977. doi: 10.1016/j.pupt.2020.101977. Epub 2020 Nov 13. PMID 33189900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, placebo-controlled, parallel group, double-blind (sponsor-open), segmental lipopolysaccharide (LPS) challenge study of GSK2798745 in healthy participants.
Pre-assignment Details: A total of 47 participants were randomized in the study. The study was terminated due to low probability of achieving a positive outcome on the primary endpoint.
Groups:
- Placebo: Participants received two tablets of placebo in the morning on Day 1. Participants then underwent segmental challenge at 2 hours after first dose wherein LPS was instilled into the right middle segment and saline control into the lingula segment of the contralateral side. The second dose of placebo was administered 10 hours after LPS and saline challenge.
- GSK2798745: Participants received two tablets of 2.4 milligrams (mg) GSK2798745 in the morning on Day 1. Participants then underwent segmental challenge at 2 hours after first dose wherein LPS was instilled into the right middle segment and saline control into the lingula segment of the contralateral side. The second dose of a single tablet of 2.4 mg GSK2798745 was administered 10 hours after LPS and saline challenge.
Period: Overall Study
Arm/Group | Placebo | GSK2798745
Started | 25 | 22
Completed | 23 | 22
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrew consent | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2798745 | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] — All Subjects Population.
  Years | 26.4 (5.07) | 27.1 (6.02) | 26.7 (5.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 22 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - White/Caucasian/European Heritage | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Baseline Adjusted Total Protein Concentration in Broncho-alveolar (BAL) Samples at 24 Hours After Segmental LPS Challenge (26 Hours Post-first Dose)
Description: Participants underwent segmental challenge to lungs, via bronchoscopy, at 2 hours after first dose of investigational medicinal product. BAL samples were taken, via bronchoscopy and total protein was measured. Baseline (2 hours) samples were taken immediately before the LPS and saline challenges, from a segment in the left lower lobe, and post-challenge samples were taken at 24 hours (26 hours post-first dose) after the LPS and saline challenges, from the challenged segments. Evaluable Population consists of all participants for whom results of the primary analysis can be determined i.e. all randomized participants who received two correct doses of study treatment, received LPS and saline segmental challenge (in contralateral lobes) and for which results of both baseline (2 hours) and LPS lobe (26 hours) BAL samples are evaluable. This population will be based on treatment the participant actually received. Median and 95% credible interval (CrI) has been presented.
Time Frame: Baseline and at 26 hours post-first dose
Population: Evaluable Population.
Measure: Median (95% Confidence Interval); unit: Milligrams per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 23 | 22
Milligrams per liter | 348.46 [285.97 to 425.67] | 318.43 [260.18 to 389.98]
Statistical Analysis 1: Comparison: Placebo vs GSK2798745; Test type: Other; Absolute Difference = -30.46, 95% CI 2-sided [-127.07 to 65.51], Standard Error of Mean 48.662 — Absolute difference (GSK2798745 - Placebo) and 95% CrI has been presented
Statistical Analysis 2: Comparison: Placebo vs GSK2798745; Test type: Other; Percentage change = 8.73, 95% CI 2-sided [-21.41 to 31.30], Standard Error of Mean 13.453 — Percentage change on GSK2798745 relative to placebo has been presented

2. Secondary Outcome: Baseline Adjusted Total Cell Count of Neutrophils in BAL Samples at 24 Hours After Segmental LPS Challenge (26 Hours Post-first Dose)
Description: Participants underwent segmental challenge to the lungs, via bronchoscopy, at 2 hours (Baseline) after the first dose of investigational medicinal product. BAL samples were taken, via bronchoscopy and total neutrophil cell count was measured. Baseline samples were taken immediately before the LPS and saline challenges, from a segment in the left lower lobe, and post-challenge samples were taken at 24 hours (26 hours post-first dose) after the LPS and saline challenges, from the challenged segments. Median and 95% CrI at indicated time point has been presented.
Time Frame: Baseline and at 26 hours post-first dose
Population: Evaluable Population.
Measure: Median (95% Confidence Interval); unit: 10^6 cells per milliliter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 23 | 22
10^6 cells per milliliter | 58.94 [42.70 to 81.42] | 54.63 [39.21 to 75.90]
Statistical Analysis 1: Comparison: Placebo vs GSK2798745; Test type: Other; Absolute Difference = -4.26, 95% CI 2-sided [-31.49 to 22.87], Standard Error of Mean 13.679 — Absolute difference (GSK2798745 - Placebo) and 95% CrI have been presented
Statistical Analysis 2: Comparison: Placebo vs GSK2798745; Test type: Other; Percentage change = 7.31, 95% CI 2-sided [-48.20 to 41.64], Standard Error of Mean 22.837 — Percentage change on GSK2798745 relative to placebo has been presented

3. Secondary Outcome: Baseline Adjusted Differential Cell Count of Neutrophils in BAL Samples at 24 Hours After Segmental LPS Challenge (26 Hours Post-first Dose)
Description: Participants underwent segmental challenge to the lungs, via bronchoscopy, at 2 hours after the first dose of investigational medicinal product. BAL samples were taken, via bronchoscopy and total neutrophil cell count was measured. Baseline samples were taken immediately before the LPS and saline challenges, from a segment in the left lower lobe, and post-challenge samples were taken at 24 hour (26 hours post-first dose) after the LPS and saline challenges, from the challenged segments. Median and 95% CrI at the indicated time point has been presented.
Time Frame: Baseline and at 26 hours post-first dose
Population: Evaluable Population.
Measure: Median (95% Confidence Interval); unit: Percentage of total cell count
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 23 | 22
Percentage of total cell count | 58.57 [54.37 to 63.09] | 58.54 [54.22 to 63.12]
Statistical Analysis 1: Comparison: Placebo vs GSK2798745; Test type: Other; Absolute Difference = -0.06, 95% CI 2-sided [-6.28 to 6.20], Standard Error of Mean 3.178 — Absolute difference (GSK2798745 - Placebo) and 95% CrI have been presented
Statistical Analysis 2: Comparison: Placebo vs GSK2798745; Test type: Other; Percentage change = 0.10, 95% CI 2-sided [-11.15 to 10.16], Standard Error of Mean 5.429 — Percentage change on GSK2798745 relative to placebo has been presented

4. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth effect and other important medical events. All Subjects Population consists of all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participant actually received. SAEs and non-SAEs were analyzed up to follow-up or early withdrawal (FU/EW) of Day 9.
Time Frame: Up to Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Participants
  Any SAE | 0 | 0
  Any non-SAE | 10 | 7

5. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters
Description: Blood samples were collected for the analysis of clinical chemistry parameters including alkaline phosphate (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST) and creatinine kinase (CK). Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
International units per liter
  ALP, Day 2 | 1.64 (8.144) | 4.00 (7.578)
  ALP, Day 9 | -3.20 (7.953) | -1.86 (6.198)
  ALT, Day 2 | 1.2 (16.87) | -3.5 (3.08)
  ALT, Day 9 | 4.4 (26.94) | -2.6 (5.14)
  AST, Day 2 | 18.4 (109.78) | -2.3 (3.97)
  AST, Day 9 | -0.2 (10.79) | -1.7 (3.83)
  CK, Day 2 | 1196.0 (6333.76) | -60.9 (59.96)
  CK, Day 9 | -239.2 (1091.86) | -37.5 (75.43)

6. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters: Direct Bilirubin, Total Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameters direct bilirubin, total bilirubin and creatinine. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Micromoles per liter
  Direct bilirubin, Day 2 | 0.8824 (0.72998) | 0.8939 (0.78261)
  Direct bilirubin, Day 9 | 0.3010 (0.85966) | 0.3187 (1.07930)
  Total bilirubin, Day 2 | 3.7552 (3.91607) | 4.2284 (4.96144)
  Total bilirubin, Day 9 | 0.0616 (5.13211) | 1.1115 (6.29042)
  Creatinine, Day 2 | -4.7029 (8.78354) | -6.4291 (8.07523)
  Creatinine, Day 9 | -4.6322 (9.99897) | -4.6611 (7.82718)

7. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters: Calcium, Glucose, Potassium, Sodium and Urea/Blood Urea Nitrogen (BUN)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including calcium, glucose, potassium, sodium and urea/BUN. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Millimoles per liter
  Calcium, Day 2 | -0.052 (0.0653) | -0.051 (0.1052)
  Calcium, Day 9 | -0.009 (0.0888) | 0.020 (0.0794)
  Glucose, Day 2 | 1.12130 (1.787201) | 0.77714 (1.785548)
  Glucose, Day 9 | -0.10214 (0.834757) | 0.06813 (0.814014)
  Potassium, Day 2 | -0.530 (0.4884) | -0.445 (0.4781)
  Potassium, Day 9 | -0.039 (0.4104) | 0.085 (0.2389)
  Sodium, Day 2 | 0.6 (2.14) | 0.9 (2.14)
  Sodium, Day 9 | 0.2 (1.82) | -0.3 (2.10)
  Urea, Day 2 | -1.1710 (1.36145) | -0.8114 (1.10273)
  Urea, Day 9 | -0.3142 (1.22512) | -0.6978 (1.21927)

8. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameter-C Reactive Protein (CRP)
Description: Blood samples were collected for the analysis of clinical chemistry parameter- CRP. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Milligrams per liter
  Day 2 | 10.98 (7.330) | 13.25 (9.186)
  Day 9 | 1.40 (2.505) | 0.92 (1.825)

9. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameter-Total Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameter- total protein. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Grams per liter
  Day 2 | -0.6 (3.50) | 0.7 (5.35)
  Day 9 | -0.6 (4.20) | 1.0 (4.57)

10. Secondary Outcome: Change From Baseline Values for Hematology Parameters
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet count and white blood cell (WBC) count. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Giga cells per liter
  Basophils, Day 2 | -0.02 (0.050) | -0.01 (0.035)
  Basophils, Day 9 | -0.01 (0.053) | 0.00 (0.044)
  Eosinophils, Day 2 | -0.01 (0.067) | -0.05 (0.118)
  Eosinophils, Day 9 | 0.01 (0.108) | -0.05 (0.106)
  Lymphocytes, Day 2 | -0.67 (0.542) | -0.40 (0.359)
  Lymphocytes, Day 9 | -0.48 (0.471) | 0.71 (4.949)
  Monocytes, Day 2 | -0.04 (0.250) | 0.04 (0.176)
  Monocytes, Day 9 | -0.04 (0.142) | -0.12 (0.123)
  Neutrophils, Day 2 | 1.18 (2.346) | 1.89 (3.083)
  Neutrophils, Day 9 | -0.94 (1.943) | -1.14 (2.418)
  Platelet count, Day 2 | -16.6 (17.63) | -15.0 (23.63)
  Platelet count, Day 9 | 6.2 (24.19) | 21.1 (22.29)
  WBC count, Day 2 | 0.42 (2.323) | 1.50 (3.071)
  WBC count, Day 9 | -1.46 (1.999) | -1.65 (2.371)

11. Secondary Outcome: Change From Baseline Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter: hemoglobin. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Grams per liter
  Day 2 | 0.1 (6.88) | 1.5 (7.25)
  Day 9 | -3.4 (6.39) | -3.6 (5.70)

12. Secondary Outcome: Change From Baseline Values for Hematology Parameters: Hematocrit and Reticulocytes
Description: Blood samples were collected for the analysis of hematology parameters: hematocrit and reticulocytes. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Percentage of red blood cells in blood
  Hematocrit, Day 2 | -0.015 (0.0228) | -0.010 (0.0213)
  Hematocrit, Day 9 | -0.025 (0.0237) | -0.027 (0.0167)
  Reticulocytes, Day 2 | -0.0000 (0.00162) | -0.0002 (0.00150)
  Reticulocytes, Day 9 | 0.0022 (0.00227) | 0.0013 (0.00247)

13. Secondary Outcome: Change From Baseline Values for Hematology Parameter: Mean Corpuscular Hemogloblin (MCH)
Description: Blood samples were collected for the analysis of hematology parameter: MCH. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Picograms
  Day 2 | 0.04 (0.300) | 0.10 (0.312)
  Day 9 | -0.02 (0.335) | 0.06 (0.357)

14. Secondary Outcome: Change From Baseline Values for Hematology Parameter: Mean Corpuscular Volume (MCV)
Description: Blood samples were collected for the analysis of hematology parameter: MCV. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Femtoliters
  Day 2 | -2.83 (2.755) | -2.59 (1.478)
  Day 9 | -2.93 (2.313) | -3.15 (1.760)

15. Secondary Outcome: Change From Baseline Values for Hematology Parameter: Red Blood Cell (RBC) Count
Description: Blood samples were collected for the analysis of hematology parameter: RBC count. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1)and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Tera cells per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Tera cells per liter
  Day 2 | -0.004 (0.2382) | 0.038 (0.2524)
  Day 9 | -0.118 (0.2221) | -0.128 (0.1929)

16. Secondary Outcome: Change From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected for measurement of urine pH at indicated time points. pH is a measure of hydrogen ion concentration and used to determine the acidity or alkalinity of urine. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
pH
  Day 2 | -0.3 (1.21) | 0.0 (1.20)
  Day 9 | -0.4 (1.12) | 0.2 (1.19)

17. Secondary Outcome: Change From Baseline in Urine Specific Gravity
Description: Urine samples were collected for the analysis of urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The dipstick test gives results in a semi-quantitative manner. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Day 2 and Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Ratio
  Day 2 | -0.0010 (0.00946) | 0.0016 (0.00836)
  Day 9 | -0.0004 (0.00721) | -0.0041 (0.00908)

18. Secondary Outcome: Number of Participants With Worst Case Post Baseline Abnormal Electrocardiogram (ECG) Findings
Description: A single 12-lead ECG was performed at the specified timepoints during the study where the participant was instructed to be in semi-recumbent position for 5 minutes before obtaining the ECG. An ECG machine that automatically calculated the heart rate and measures like the PR, QRS, QT, and corrected QT intervals. Number of participants with worst-case post-Baseline abnormal clinically significant findings and abnormal not clinically significant findings in ECG results has been reported. The decision if an ECG abnormality is clinically significant or not-clinically significant was in the discretion of the investigator, based on her/his clinical judgement. Baseline values is defined as the latest pre-treatment assessment with a non-missing value.
Time Frame: Up to Day 9 (FU/EW)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Participants
  Abnormal-not clinically significant | 21 | 20
  Abnormal-clinically significant | 0 | 0

19. Secondary Outcome: Number of Participants With Abnormal Findings During Physical Examinations
Description: A complete physical examination included, at a minimum, assessments of the skin, cardiovascular, respiratory, gastrointestinal and neurological systems. Height and weight were also measured and recorded. A brief physical examination included, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen).
Time Frame: Up to Day 9 (FU/EW)
Population: Safety Population. This analysis was not planned and data was not collected and captured in the database.
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: The DBP and SBP were measured in participants in a semi-supine position after 5 minutes rest. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 1, 6, 12, 14, 30 hours and Day 9 (FU/EW)
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Millimeters of mercury
  DBP, 1 hour, n=25, 22 | 1.34 (4.945) | -1.34 (4.568)
  DBP, 6 hours, n=25, 22 | 2.46 (5.006) | 4.25 (5.642)
  DBP, 12 hours, n=25, 22 | 3.70 (4.409) | -0.07 (7.053)
  DBP, 14 hours, n=24, 22: number analyzed (Participants) | 24 | 22
  DBP, 14 hours, n=24, 22 | 2.77 (6.694) | 0.43 (6.225)
  DBP, 30 hours, n=25, 22 | 1.86 (5.088) | 1.75 (5.026)
  DBP, Day 9, n=25, 22 | -0.06 (6.009) | -0.70 (5.719)
  SBP, 1 hour, n=25, 22 | -1.20 (6.722) | 1.07 (8.839)
  SBP, 6 hours, n=25, 22 | 6.92 (6.372) | 7.30 (7.428)
  SBP, 12 hours, n=25, 22 | 8.64 (5.959) | 5.66 (9.713)
  SBP, 14 hours, n=24, 22: number analyzed (Participants) | 24 | 22
  SBP, 14 hours, n=24, 22 | 8.35 (8.098) | 4.84 (7.078)
  SBP, 30 hours, n=25, 22 | 7.20 (5.681) | 5.02 (9.380)
  SBP, Day 9, n=25, 22 | 2.48 (7.913) | -0.98 (8.574)

21. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured at indicated time points in supine position after 5 minutes rest for the participants. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 1, 6, 12, 14, 30 hours and Day 9 (FU/EW)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Beats per minute
  1 hour, n=25, 22 | -3.28 (7.666) | -3.61 (11.640)
  6 hours, n=25, 22 | 13.12 (8.402) | 11.75 (11.732)
  12 hours, n=25, 22 | 14.56 (11.438) | 11.89 (13.917)
  14 hours, n=24, 22: number analyzed (Participants) | 24 | 22
  14 hours, n=24, 22 | 14.00 (13.808) | 11.84 (14.937)
  30 hours, n=25, 22 | 14.40 (11.183) | 17.02 (10.239)
  Day 9, n=25, 22 | 1.44 (8.885) | -1.02 (9.749)

22. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature was measured at indicated time points in supine position after 5 minutes rest for the participants. Baseline values were defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 1, 2, 6, 8, 12, 14, 30 hours and Day 9 (FU/EW)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Degree celsius
  1 hour, n=25, 22 | -0.06 (0.380) | 0.01 (0.256)
  2 hours, n=25, 22 | -0.22 (0.485) | -0.06 (0.362)
  6 hours, n=25, 22 | 0.09 (0.411) | 0.07 (0.400)
  8 hours, n=25, 22 | 0.12 (0.473) | 0.21 (0.537)
  12 hours, n=25, 22 | 0.65 (0.395) | 0.74 (0.735)
  14 hours, n=24, 22: number analyzed (Participants) | 24 | 22
  14 hours, n=24, 22 | 0.63 (0.523) | 0.84 (0.764)
  30 hours, n=25, 22 | 0.10 (0.434) | 0.26 (0.286)
  Day 9, n=25, 22 | -0.20 (0.612) | -0.11 (0.803)

23. Secondary Outcome: Number of Participants With Positive Fecal Occult Blood Test (FOBT) Data
Description: Based on the preclinical finding of gastric erosions, FOBT was performed before and after dosing at screening and follow-up and any positive hemoglobin measurement was recorded as potentially clinically important. Participants with at least one recorded result has been reported.
Time Frame: At Day 9
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Participants | 0 | 1

24. Secondary Outcome: Mean Forced Expiratory Volume in 1 Second (FEV1) and Mean Forced Vital Capacity (FVC)
Description: Spirometric assessments including FEV1 and FVC were conducted from screening and up to Day 9. Measurements were made in triplicate and the highest FEV1 and FVC were recorded in the case report form (CRF). Mean FEV1 and FVC values along with 95% confidence interval (CI) at indicated timepoints has been presented. Baseline values is defined as the latest pre-treatment assessment with a non-missing value.
Time Frame: Baseline (Day 1, Pre-dose) pre-bronchodilator and at Day 1 (pre-bronchodilator and 6 Hours), at Day 2 (25.5 and 30 Hours) and Day 9 pre-bronchodilator
Population: as for outcome 20
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 25 | 22
Liters
  FEV1, Day 1, Pre-bronchodilator, n=25, 22 | 4.651 [4.352 to 4.950] | 4.744 [4.491 to 4.997]
  FEV1, Day 1, 6 Hours, n=25, 22 | 4.564 [4.268 to 4.860] | 4.658 [4.396 to 4.920]
  FEV1, Day 2, 25.5 Hours, n=23, 22: number analyzed (Participants) | 23 | 22
  FEV1, Day 2, 25.5 Hours, n=23, 22 | 4.496 [4.233 to 4.759] | 4.704 [4.433 to 4.975]
  FEV1, Day 2, 30 Hours, n=23, 22: number analyzed (Participants) | 23 | 22
  FEV1, Day 2, 30 Hours, n=23, 22 | 4.419 [4.147 to 4.691] | 4.617 [4.326 to 4.909]
  FEV1, Day 9, pre-bronchodilator, n=25, 22 | 4.640 [4.346 to 4.935] | 4.796 [4.517 to 5.075]
  FVC, Day 1, Pre-bronchodilator, n=25, 22 | 5.834 [5.516 to 6.153] | 5.867 [5.544 to 6.190]
  FVC, Day 1, 6 Hours, n=25, 22 | 5.647 [5.316 to 5.978] | 5.711 [5.372 to 6.051]
  FVC, Day 2, 25.5 Hours, n=23, 22: number analyzed (Participants) | 23 | 22
  FVC, Day 2, 25.5 Hours, n=23, 22 | 5.699 [5.392 to 6.006] | 5.820 [5.467 to 6.172]
  FVC, Day 2, 30 Hours, n=23, 22: number analyzed (Participants) | 23 | 22
  FVC, Day 2, 30 Hours, n=23, 22 | 5.497 [5.189 to 5.806] | 5.642 [5.281 to 6.002]
  FVC, Day 9, pre-bronchodilator, n=25, 22 | 5.769 [5.453 to 6.085] | 5.863 [5.513 to 6.214]

25. Secondary Outcome: Area Under the Curve During 26 Hours of GSK2798745
Description: Blood samples were collected at indicated time points. The 2 and 26-hour blood samples were taken immediately before BAL sampling. Pharmacokinetic (PK) Population consists of all participants in the All Subjects Population who had at least one non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 6, 8, 12, 12.5, 13, 13.5, 14, 15, 24 and 26 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | GSK2798745
Number analyzed (Participants) | 22
Hour*nanograms per milliliter | 221.27 (20.8)

26. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK2798745
Description: Blood samples were collected at indicated time points. The 2- and 26-hour blood samples were taken immediately before BAL sampling.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 6, 8, 12, 12.5, 13, 13.5, 14, 15, 24 and 26 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | GSK2798745
Number analyzed (Participants) | 22
Nanograms per milliliter | 14.821 (17.7)

ADVERSE EVENTS:
Time Frame: SAEs and non-SAEs were collected up to Day 9.
Description: SAEs and non-SAEs were summarized for All Subjects Population
Arm/Group | Placebo | GSK2798745
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22
Other Adverse Events (participants affected / at risk) | 10/25 | 7/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | GSK2798745 (N=22)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Pyrexia (General disorders) | 3 (3) | 4 (5)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT03511105/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT03511105/SAP_001.pdf